CLINICAL TRIAL: NCT01732523
Title: Predictive Value of Carotid Lesion Neovascularization Detected by Contrast-enhanced Ultrasound (CEUS) in Patients With Asymptomatic Carotid Stenosis
Brief Title: Predictive Value of Neovascularization Within Asymptomatic Carotis Stenosis on CEUS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EK145/12; PZ00P3_142419/1 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2012-11-16; First posted 2012-11-26 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Carotid Stenosis
Keywords: Carotid stenosis; Vasa Vasorum; Ultrasonography
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No treatment: No intervention
  Interventions: Diagnostic Test: Contrast enhanced carotid ultrasound

INTERVENTIONS:
Diagnostic Test: Contrast enhanced carotid ultrasound

SUMMARY:
Atherosclerosis is a chronic, systemic and progressive disease affecting different arterial blood vessels in the body. Atherosclerotic lesions silently progress from small plaques to severe stenosis and may remain asymptomatic for years. Unstable plaques and stenosis (also called vulnerable plaques), however, are prone to rupture leading to myocardial infarction, or stroke. The proliferation of the small arteries that are distributed to the outer and middle coats of the larger blood vessels (vasa vasorum) and within the atherosclerotic plaques (neovascularization) are inherently linked with the atherosclerotic plaque development, plaque inflammation and vulnerability. By injecting ultrasound contrast agents (microbubbles) into the blood stream, it is possible to detect this microcirculation of the vessel wall and the neovascularization within the atherosclerotic plaque using a contrast-enhanced ultrasound (CEUS) imaging technique. Particularly, CEUS of the carotid artery has been introduced as a non-invasive technique to improve detection of carotid atherosclerosis and to evaluate the presence of carotid plaque neovascularization which has emerged as a new marker for plaque vulnerability. The project investigates the predictive value of the detection of carotid plaque neovascularization on CEUS imaging in patients with asymptomatic carotid artery stenosis regarding the progression of the carotid atherosclerotic lesion and future vascular events including myocardial infarction, stroke or vascular intervention. The investigators hypothesize that neovascularization within the carotid lesion will significantly be more pronounced in patients with progressive carotid lesions and in patients suffering future vascular events during. The project will support the concept that intraplaque neovascularization is associated with plaque instability and vulnerability and therefore, the use of CEUS may provide an additional non-invasive, simple, safe, and reliable imaging modality to risk stratify individuals. The identification of vulnerable that are at increased risk of rupture by identification of intraplaque neovascularization is expected to improve the prediction of future vascular events and thus allow for better treatment selection. It will help the clinician to further risk stratify carotid stenosis. Particularly, it will help to identify unstable carotid stenosis that may already benefit from invasive therapy as carotid thromboendarterectomy and stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients age > 18 years
* Asymptomatic (no history of cerebrovascular event in the corresponding vessel territory) ≥30% carotid stenosis on standard carotid ultrasound

Exclusion Criteria:

* History of previous carotid endarterectomy or carotid stenting.
* Heart failure (HYHA III or IV)
* Myocardial infarction (<7d)
* Severe pulmonal-arterial hypertension (pulmonal arterial pressure >90mmHg) based on clinical information (history of pulmonal arterial pressure, dyspnea on exertion New York Heart Association (NYHA) III and NYHA IV)
* pregnancy (pregnancy test in patients of childbearing age: <50 years and/or less than 2 years after menopause)
* Follow-up is not considered feasible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In-and out-patients referred to our ultrasound laboratory for carotid ultrasound for a clinical indication (preoperative, carotid murmur, known carotid lesion) will be ask to participate in this clinical study and will be asked to undergo study carotid ultrasound including CEUS.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Vascular event or vascular intervention | 10 years
  The endpoint assessed will be the occurrence of any vascular event or vascular intervention. This composite end point includes any death of presumed vascular origin (fatal stroke, fatal myocardial infarction, sudden death, other vascular death), nonfatal stroke and TIA, nonfatal myocardial infarction, and any arterial vascular intervention that had not already been planned at the time of inclusion (eg, carotid surgery or angioplasty/stenting, coronary bypass, percutaneous coronary intervention, peripheral vascular surgery or angioplasty/stenting). All events and vascular interventions should be confirmed by hospital discharge report and medical files.

SECONDARY OUTCOMES:
Progression of carotid stenosis over time | 10 years
  progression of carotid stenosis over time (progression in the lesion area, lesion volume, and degree of stenosis) assessed by yearly repeated standard carotid ultrasound study. Based on the yearly repeated standard carotid ultrasound studies progression rate of the lesion area and the lesion volume can be quantified for each stenosis and specify as continuous variable in cm2/year (area progression/year) and in cm3/year (volume progression/year). Additionally, the progression of the grade of stenosis will be quantified as categorical variable by determining the change of the stenosis category over time (30-49%, 50-69%, 70-99%, 100%) (Stable stenosis or increase in 1, 2, or 3 categories over 5 years).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Staub, MD, Principal Investigator — University Hospital Basle, Angiology
Locations (1):
- Unversity Hospital Basel, Angiology, Basel, Switzerland